CLINICAL TRIAL: NCT02215733
Title: The Use of Angiotensin Receptor Blockers and the Risk of Cancer
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 502.599
Record Dates: First submitted 2014-08-12; First posted 2014-08-13 (Estimated); Last update posted 2014-08-13 (Estimated); Status verified 2014-08

CONDITIONS: Neoplasm
MeSH Terms: conditions — Neoplasms | interventions — Adrenergic beta-Antagonists; Diuretics; Telmisartan

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- Patients prescribed antihypertensives
  Interventions: Drug: ARB; Drug: ACEI; Drug: Beta-blockers; Drug: Diuretics; Drug: Telmisartan

INTERVENTIONS:
Drug: ARB — other than telmisartan
Drug: ACEI
Drug: Beta-blockers
Drug: Diuretics
Drug: Telmisartan

SUMMARY:
The primary objective of this study was to assess whether angiotensin blockers (ARBs) and telmisartan in particular, are associated with an increased overall risk of the four most common cancers, namely, lung, colorectal, breast and prostate cancers. A secondary objective was to explore these effects separately for each of the four cancers and in combination with angiotensin-converting-enzyme-inhibitors (ACEIs).

ELIGIBILITY:
Inclusion Criteria:

* Patients prescribed an antihypertensive agent between 01-JAN-1995 and 31-DEC-2008 with at least two years of up-to-standard medical history in United Kingdom's General Practice Research Database (GPRD)

Exclusion Criteria:

* History of cancer at any time prior to cohort entry

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients prescribed an antihypertensive agent between January 1, 1995 and December 31, 2008, with follow-up until December 31, 2010 Information extracted from United Kingdom General Practice Research Database (GPRD)
Sampling Method: Probability Sample
Enrollment: 1165781 (Actual)
Dates: Start 2011-02; Primary Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Number of patients with occurrences of lung, colorectal, breast and prostate cancers related to use of ARBs | 16 years
Determination of dose-response in terms of ARB duration of use and cumulative dose and the risk of lung, colorectal, breast and prostate cancers combined | 16 years
Ratio of occurrence of lung, colorectal, breast and prostate cancers related to use of ARBs, relative to beta-blockers and diuretics | 16 years
Ratio of occurrence of lung, colorectal, breast and prostate cancers related to use of telmisartan, relative to beta-blockers and diuretics | 16 years
Ratio of occurrence of lung, colorectal, breast and prostate cancers related to use of telmisartan relative to other ARBs | 16 years

SECONDARY OUTCOMES:
Number of patients with occurrences of lung cancer related to use of ARBs alone | 16 years
Number of patients with occurrences of colorectal cancer related to use of ARBs alone | 16 years
Number of patients with occurrences of breast cancer related to use of ARBs alone | 16 years
Number of patients with occurrences of prostate cancer related to use of ARBs alone | 16 years
Number of patients with occurrences of lung cancer related to use of ARBs with ACEI | 16 years
Number of patients with occurrences of colorectal cancer related to use of ARBs with ACEI | 16 years
Number of patients with occurrences of breast cancer related to use of ARBs with ACEI | 16 years
Number of patients with occurrences of prostate cancer related to use of ARBs with ACEI | 16 years
Ratio of occurrence of lung cancer related to use of telmisartan relative to other ARBs | 16 years
Ratio of occurrence of colorectal cancer related to use of telmisartan relative to other ARBs | 16 years
Ratio of occurrence of breast cancer related to use of telmisartan relative to other ARBs | 16 years
Ratio of occurrence of prostate cancer related to use of telmisartan relative to other ARBs | 16 years